CLINICAL TRIAL: NCT06034275
Title: An Open-label, Multicenter Phase 1 Study to Characterize Safety, Tolerability, Preliminary Antitumor Activity, Pharmacokinetics, and Pharmacodynamics of VIP943 Monotherapy in Subjects With Advanced CD123+ Hematologic Malignancies
Brief Title: Study of VIP943 in Subjects With Advanced CD123+ Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vincerx Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VNC-943-101
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia; B-cell Acute Lymphoblastic Leukemia; High-risk Myelodysplastic Syndrome
Keywords: ADC; Hematologic Malignancies; Leukemia; CD123; B-ALL; AML; MDS; Relapsed/ Refractory; Hematologic Diseases; Bone Marrow Diseases
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hematologic Neoplasms; Leukemia; Hematologic Diseases; Bone Marrow Diseases

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation of VIP943 (QW) (Experimental): Subjects with AML, MDS, and B-ALL with CD123 expression will be administered VIP 943 in sequential ascending doses as a monotherapy via intravenous (IV) administration weekly (QW).
  Interventions: Drug: VIP943 (QW)
- Dose Escalation of VIP943 (BIW) (Experimental): Subjects with AML, MDS, and B-ALL with CD123 expression will be administered VIP 943 in sequential ascending doses as a monotherapy via intravenous (IV) administration twice weekly (BIW).
  Interventions: Drug: VIP943 (BIW)

INTERVENTIONS:
Drug: VIP943 (QW) — VIP943 will be administered by IV Infusion weekly
  Arms: Dose Escalation of VIP943 (QW)
Drug: VIP943 (BIW) — VIP943 will be administered by IV Infusion bi-weekly
  Arms: Dose Escalation of VIP943 (BIW)

SUMMARY:
Dose Escalation - Determine the maximum tolerated dose (MTD), if possible, or minimum optimal biologic dose (OBD), and evaluate the safety and tolerability of VIP943 in subjects with advanced CD123+ hematologic malignancies

DETAILED DESCRIPTION:
Relapsed or refractory AML, MDS, or B-ALL subjects who are CD123 positive. Subjects must have exhausted all available standard therapies or be deemed ineligible for potential available therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed AML, B-ALL or MDS. Subjects must have exhausted all available standard therapies or be deemed ineligible for potential available therapies.
* Evidence of ≥5% bone marrow or blood blasts (acute leukemia) or ≥5% bone marrow or blood myeloblasts (MDS) to allow for assessment of drug activity.
* Evidence of CD123 expression from a local laboratory.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2

Exclusion Criteria:

* Known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Clinically significant cardiac disease including congestive heart failure > New York Heart Association (NYHA) Class II), evidence for coronary artery disease (eg, unstable angina (anginal symptoms at rest) or new-onset angina (within the last 6 months or myocardial infarction within the past 6 months before first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT (Dose limit toxicity) of VIP943 | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 28 days

SECONDARY OUTCOMES:
Response rate to VIP943 as assessed by investigators using disease-specific response criteria | Cycle 1 Day 1 up to 30 days after the last dose, where each cycle is up to 28 days (up to approximately 10 months)
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) of VIP943 | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 28 days
Area under the concentration versus time curve from zero to infinity after single (first) dose (AUC) of VIP943 | Cycle 1 Day 1 through Cycle 2 Day 1, where each cycle is up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Vincerx Study Director, Study Director — Vincerx Pharma, Inc.
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Cincinnati, Cincinnati, Ohio
  - TriStar Bone Marrow Transplant, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No